CLINICAL TRIAL: NCT07361913
Title: A Multicentre, Randomised Cross-over Equivalence Trial Investigating Knowledge of Anatomy Following Virtual Reality or Standard Teaching in Novice Anaesthetists
Brief Title: RA Anatomy - VRvST Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal National Orthopaedic Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: WKR0-2024-0032; IRAS Project ID: 356761 (Other: HRA and Health and Care Research Wales (HCRW))
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-10

CONDITIONS: Virtual Reality Simulation; Virtual Reality; Education, Medical
Keywords: Virtual reality; sonoanatomy; regional anaesthesia

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard teaching (Active Comparator): Standard anatomical training
  Interventions: Other: Standard anatomy model teaching
- Virtual reality (Experimental): Virtual reality based anatomical training
  Interventions: Other: 3D virtual reality anatomy teaching

INTERVENTIONS:
Other: 3D virtual reality anatomy teaching — Knowledge of regional nerve anatomy among novice anaesthetists using 3D virtual reality is equivalent to standard teaching
  Arms: Virtual reality
Other: Standard anatomy model teaching — Knowledge of regional nerve anatomy among novice anaesthetists using standard anatomy model teaching
  Arms: Standard teaching

SUMMARY:
Primary Objective: Score out of 44 on a validated test of anatomy and sono-anatomy

Secondary Objective:

Before training

* Handedness (Edinburgh Handedness Inventory)
* Subjective sleepiness (Karolinska scale)
* Motor reaction time (Psychomotor Vigilance test)
* Attention control (Anti-Saccade test)
* Mental rotation (Mental Rotation Task)
* Depression Anxiety, Stress (DASS score)
* Visual Search Task (Divided Attention)
* Knowledge pretraining

After training and testing

* Knowledge after training session
* Acceptability: Client Satisfaction Questionnaire (CSQ-8)
* Usability: CyberSickness in Virtual Reality Questionnaire (CSQ-VR)
* Immersion: Witmer and Singer Presence Questionnaire
* Subjective workload (NASA - TLX scale)
* Cognitive Demand Battery (CBD)
* Resource use: Calculation of cost differences between learning Modalities

Study population: Resident anaesthetists

Recruitment Target: 102

Methodology:

This is a non-clinical randomised controlled trial of resident anaesthetists undergoing training in regional anaesthesia. Residents will be randomised to one of two groups for each training session day:

* Standard anatomical training (Group A)
* Virtual reality based anatomical training. (Group B) Then followed by another training day session and participants will enter either standard or VR teaching depending on the previous allocation:
* Standard anatomical training (Group B)
* Virtual reality based anatomical training. (Group A)

Anatomical knowledge will be tested in both groups using an on-line questionnaire developed by the Chief Investigator.

Eligibility criteria: Inclusion criteria:

1. Anaesthetists that are residents in a recognised Royal College of Anaesthetists (RCoA) training program
2. Anaesthetic training grades (Stage 1 - 3).

Exclusion criteria:

1. Visual impairment (this does not include wearing glasses/contact lenses)
2. History of severe diseases affecting physical motion or balance
3. History of any drugs that may affect physical motion or balance within 12 hours of the intervention
4. Pregnancy
5. Individuals who had consumed alcohol within 24 h of the intervention.
6. Resident doctors not in a recognised RCOA training program e.g. Staff grade anaesthetists.

Study treatment:

Standard teaching - control Virtual reality teaching - intervention

DETAILED DESCRIPTION:
STUDY RATIONALE AND RISK/BENEFIT ANALYSIS We propose that in order to develop a sound knowledge of anatomy and sono-antomy, virtual reality could be used as an aid to understanding and interpreting 2-D sono-antomical structures. Trainees will have an enhanced learning experience that reinforces the skills required to perform safe regional anaesthesia.

Hypothesis: We hypothesise that knowledge of regional nerve anatomy among novice anaesthetists using 3D virtual reality is equivalent to standard teaching.

MANAGEMENT OF POTENTIAL STUDY RISKS One potential major weakness is the risk of trainer bias when delivering training. The knowledge test was written by Dr Bellew, and that Dr Bellew and Prof McLeod will be delivering the 'VR training' and 'standard training' arms respectively. The possibility exists for the trainers to bias results by providing test-specific training to one arm, but not the other. To mitigate this risk training packages with specific anatomical areas taught and check lists will be used by an observer to ensure all aspects are taught and/or omitted as per the training package.

Virtual reality is usually regarded as safe to use. There are reports of it causing headache, eyestrain, fatigue, blurred vision and dizziness with prolonged use. These symptoms tend to get better shortly after participants stop using the virtual reality equipment. We will minimise the risk of these symptoms by limiting the use of the virtual reality headset to 2 - 3 x 30-40 minute sessions within an eight-hour period. We will be assessing for these side effects using validated questionnaires. Also, the VR environment will be projected onto a screen for participants if they need to remove the VR equipment.

PRIMARY OBJECTIVE Our primary aim is to study knowledge of anatomy following initial VR teaching compared to standard teaching.

Primary end-point: Score out of 44 on a validated test of anatomy and sono-anatomy

SECONDARY OBJECTIVES

Secondary objectives and end-points:

Before training

* Handedness (Edinburgh Handedness Inventory)
* Subjective sleepiness (Karolinska scale)
* Motor reaction time (Psychomotor Vigilance test)
* Attention control (Anti-Saccade test)
* Mental rotation (Mental Rotation Task)
* Depression Anxiety, Stress (DASS score)
* Visual Search Task (Divided Attention)
* Knowledge pretraining After training and testing
* Knowledge after each training session
* Acceptability: Client Satisfaction Questionnaire (CSQ-8)
* Usability: CyberSickness in Virtual Reality Questionnaire (CSQ-VR)
* Immersion: Witmer and Singer Presence Questionnaire
* Subjective workload (NASA - TLX scale)
* Cognitive Demand Battery (CBD)
* Resource use: Calculation of cost differences between learning modalities

Experimental design and methods (Workpackage (WP); Milestone (M); Deliverables (D)) WP 1 Baseline measurements M 1.1 Confirmation of capacity and capability (C&C) at each site M 1.2 Inclusion criteria: anaesthetists (non-pregnant) from London, Nottingham, Tayside, Sunderland.

M 1.3 Measure online participant characteristics and psychometric measures (secondary outcomes as above) using web based Inquisit Lab 5 platform (Millisecond Software, Seattle).

D1 Report results. WP 2 Training and testing M 2.1 Randomisation Participants will be randomised to one of two groups

* Standard training
* VR based training M 2.2 Psychometric testing (pre training secondary end points as above) M 2.3 VR familiarisation VR training will be preceded by VR familiarisation. Participants will wear Meta Quest 3 VR glasses and learn upper and lower limb anatomy using the 3D Organon package https://www.3dorganon.com/ that also incorporates sono-anatomy related to regional anaesthesia M 2.4 Training will be structured, last 30 - 40 min and follow the principles of deliberate practice. Training will consist of 1:1 trainer: trainee interaction with feedback either after the VR session or during the standard training session.

Training will cover upper and lower limb blocks, truncal and abdominal blocks. The standard session will consist of a lecture followed by learning on a plastic anatomical model. All training to be provided by Dr Bellew and Prof McLeod at all centres M 2.5 Testing Knowledge will be tested four occasions and pseudoanonymised using a random code generator.

* Before training
* After training M 2.6 Questionnaire feedback
* Post-test secondary endpoints as above D 2.1 Conference paper D 2.2 Journal submission Testing consists of questions involving sono-anatomy video clips of nerve blocks. The tests will be completed on the on-line platform (r)14 with a built in time limit. Answers will be free-text and marked by two blinded raters. All participants will be allocated a code so that results could be pseudo-anonymised.

INCLUSION CRITERIA Anaesthetists that are in a recognised Royal College of Anaesthetists (RCoA) training program in the Uk, Anaesthetic training grades (Stage 1 - 3).

EXCLUSION CRITERIA

* Visual impairment (this does not include wearing glasses/contact lenses)
* History of severe diseases affecting physical motion or balance
* History of any drugs that may affect physical motion or balance within 12 hours of the intervention
* Pregnancy
* Individuals who had consumed alcohol within 24 h of the intervention.

PARTICIPANT RECRUITMENT PROCESS

Participant recruitment at a site will only commence once the study team has ensured that the following approvals/essential documents are in place:

1. Health Research Authority (HRA) approval
2. Local Site Delegation of Duties and Signature Log is completed (if applicable)
3. Confirmation of Capacity and Capability.

All sites participating in the study will also be asked to provide a copy of the following:

1. Signed Organisation Information Document (OID) or model agreement, as agreed with the Sponsor
2. Confirmation of Capacity and Capability
3. Sponsor greenlight (if applicable). Potential participants will be those resident doctors enrolled in a RCoA recognised anaesthetic training program. Participants will be recruited via advertised email to anaesthetic departments in the UK, Heads of Schools of training will also be asked to disseminate emails and via local messaging groups within the various Schools of anaesthesia.

INFORMED CONSENT Consent to enter the study will be sought from each participant only after a full explanation has been given, an information leaflet offered, and time allowed for consideration. Signed participant consent will be obtained. The right of the participant to refuse to participate without giving reasons must be respected. All participants are free to withdraw at any time.

Informed consent will be obtained by the Chief Investigator (CI), Principal Investigator (PI) and/or a nominated deputy as recorded on Sponsor's Delegation of Responsibilities Log locally.

Consent to enter this study will be obtained after a full account has been provided of its nature, purpose, risks, burdens and potential benefits, and the participant has had the opportunity to deliberate. The participant will be allowed to specify the time they wish to spend deliberating, usually up to 24 hours.

Periods shorter than 24 hours will be permitted if the participant feels that further deliberation will not lead to a change in their decision, and provided the person seeking consent is satisfied that the participant has fully retained, understood and deliberated on the information given.

Likewise, periods longer than 24 hours will be permitted should the participant request this. The Investigator or designee will explain that the participants are under no obligation to enter the study and that they can withdraw at any time during the study, without having to give a reason.

A copy of the signed Informed Consent Form (ICF), along with a copy of the most recent approved Participant Information Sheet (PIS) will be given to the study participant. The original signed consent form will be retained at the study site and filed in the Site Investigator File (ISF) / Trial Master File (TMF).

If new safety information results in significant changes to the risk-benefit assessment, the consent form and Participant Information Sheet will be reviewed and updated if necessary. All subjects, including those already enrolled, will be informed of the new information, given a copy of the revised consent form and PIS and asked to re-consent if they choose to continue in the study.

RANDOMISATION PROCEDURE A computer-generated program for random numbers will be used for simple randomization of participants https://www.randomizer.org/

This is a non-clinical randomised controlled trial of resident anaesthetists undergoing simulation training in regional anaesthesia. Residents will be randomised to one of two groups for each training session day:

* Standard anatomical training (Group A)
* Virtual reality based anatomical training. (Group B) AND followed 2 - 4 weeks later
* Standard anatomical training (Group B)
* Virtual reality based anatomical training. (Group A)

DATA HANDLING AND ANALYSIS We will use RStudio to analyse data with appropriate packages. Examples include: Library (here, janitor, tidyverse, psych, dplyr, Hmisc, finalfit, ltm, lme4). Data will be stored on a University of Dundee managed laptop and OneDrive UoD database. Professor McLeod will be responsible for data analysis and storage. He will provide a report using Quatro.

ELIGIBILITY:
Inclusion Criteria:

* Anaesthetists that are residents in a recognised Royal College of Anaesthetists (RCoA) training program
* Anaesthetic training grades (Stage 1 - 3).

Exclusion Criteria:

* Visual impairment (this does not include wearing glasses/contact lenses)
* History of severe diseases affecting physical motion or balance
* History of any drugs that may affect physical motion or balance within 12 hours of the intervention
* Pregnancy
* Individuals who had consumed alcohol within 24 h of the intervention.
* Resident doctors not in a recognised RCOA training program e.g. Staff grade anaesthetists

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Score out of 44 on a validated test of anatomy and sono-anatomy | From enrolement to end of study day 2
  Sonoanatomy knowledge using Virtual Reality

SECONDARY OUTCOMES:
Handedness (Edinburgh Handedness Inventory) | 2 - 4 weeks prior to study day 1
Visual Search Task (Divided Attention) | 2 - 4 weeks prior to study day 1

CONTACTS AND LOCATIONS:
Overall Officials: Boyne Bellew, Principal Investigator — Royal National Orthopaedic Hospital NHS Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Motter BC, Simoni DA. Changes in the functional visual field during search with and without eye movements. Vision Res. 2008 Oct;48(22):2382-93. doi: 10.1016/j.visres.2008.07.020. Epub 2008 Sep 14. PMID 18722398
- [Background] Shepard S, Metzler D. Mental rotation: effects of dimensionality of objects and type of task. J Exp Psychol Hum Percept Perform. 1988 Feb;14(1):3-11. PMID 2964504
- [Background] Sereno AB, Holzman PS. Antisaccades and smooth pursuit eye movements in schizophrenia. Biol Psychiatry. 1995 Mar 15;37(6):394-401. doi: 10.1016/0006-3223(94)00127-O. PMID 7772648
- [Background] Thomann J, Baumann CR, Landolt HP, Werth E. Psychomotor vigilance task demonstrates impaired vigilance in disorders with excessive daytime sleepiness. J Clin Sleep Med. 2014 Sep 15;10(9):1019-24. doi: 10.5664/jcsm.4042. PMID 25142762
- [Background] Zhao J, Xu X, Jiang H, Ding Y. The effectiveness of virtual reality-based technology on anatomy teaching: a meta-analysis of randomized controlled studies. BMC Med Educ. 2020 Apr 25;20(1):127. doi: 10.1186/s12909-020-1994-z. PMID 32334594
- [Background] Chytas D, Piagkou M, Demesticha T, Tsakotos G, Natsis K. Are extended reality technologies (ERTs) more effective than traditional anatomy education methods? Surg Radiol Anat. 2022 Sep;44(9):1215-1218. doi: 10.1007/s00276-022-02998-5. Epub 2022 Aug 11. PMID 35951086
- [Background] Mathew RK; Immersive Healthcare Collaboration; Mushtaq F. Three principles for the progress of immersive technologies in healthcare training and education. BMJ Simul Technol Enhanc Learn. 2021 May 25;7(5):459-460. doi: 10.1136/bmjstel-2021-000881. eCollection 2021. No abstract available. PMID 35515725
- [Background] Orser BA, Spadafora SM. Competence-Based Training and Immersion Virtual Reality: Paradigm-Shifting Advances in Medical Education. Anesth Analg. 2022 Aug 1;135(2):220-222. doi: 10.1213/ANE.0000000000006116. Epub 2022 Jul 5. No abstract available. PMID 35839491
- See also: 2021 Anaesthetics curriculum — https://www.rcoa.ac.uk/training-careers/training-hub/2021-anaesthetics-curriculum

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-18): https://cdn.clinicaltrials.gov/large-docs/13/NCT07361913/Prot_SAP_000.pdf